CLINICAL TRIAL: NCT06389760
Title: Nimotuzumab Combined With mFOLFIRINOX/GX as Postoperative Adjuvant Therapy in Pancreatic Cancer: a Prospective, Multicenter, Single-arm, Open-label Study
Brief Title: Nimotuzumab Combined With mFOLFIRINOX/GX as Postoperative Adjuvant Therapy in Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-Nim-PC-16
Record Dates: First submitted 2024-04-11; First posted 2024-04-29 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Cancer
Keywords: Nimotuzumab; mFOLFIRINOX; adjuvant therapy; pancreatic cancer; GX
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab+ mFOLFIRINOX/GX (Experimental): Patients will receive chemotherapy (either mFOLFIRINOX or GX) plus Nimotuzumab as postoperative adjuvant therapy.
  Interventions: Drug: Nimotuzumab; Drug: mFOLFIRINOX; Drug: GX

INTERVENTIONS:
Drug: Nimotuzumab — When combined with the mFOLFIRINOX regimen, nimotuzumab (nimo) will be administered at a dose of 400mg on Day 1 and 15 of a 28-day cycle (6 cycles). When combined with the GX regimen, nimotuzumab will be given at 400mg on Day 1 and 8 of a 21-day cycle (8 cycles).
  Other Names: Taixinsheng
Drug: mFOLFIRINOX — Patients will receive mFOLFIRINOX as follows: Oxaliplatin 65 mg/m2 on Day 1 and 15 of a 28-day cycle; Irinotecan 130 mg/m2 on Day 1 and 15 of a 28-day cycle; Leucovorin(LV) 200 mg/m2 Day 1 and 15 of a 28-day cycle; 5-Fluorouracil 2.4g/m2 for 46 hours continuous infusion on Day 1 and 15 of a 28-day cycle (6 cycles).
Drug: GX — Patients will receive GX regimen as follows: Gemcitabine 1000 mg/m2 on Day 1 and 8 of a 21-day cycle; capecitabine 2000 mg/m2 on d1-14 a 21-day cycle(8 cycles).

SUMMARY:
This is a prospective, multicenter, single-arm, open-label study. The main purpose of the study is to evaluate the efficacy and safety of Nimotuzumab combined with mFOLFIRINOX/GX for postoperative adjuvant treatment of pancreatic cancer.

DETAILED DESCRIPTION:
This clinical study is designed as a prospective, multicenter, single arm, open-label study to evaluate the clinical efficacy and safety of combination Nimotuzumab with mFOLFIRINOX/GX as postoperative adjuvant therapy in pancreatic cancer. The main endpoint is disease-free survival (DFS). Additional end points included overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 years or older, gender unlimited;
* 2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* 3. Had undergone complete macroscopic resection for pancreatic cancer (R0 or R1 resection) with histological confirmation and with no evidence of distant metastasis as demonstrated by imaging;
* 4. No prior tumor therapy;
* 5. Adequate organ and bone marrow function, defined as follows: White blood cells (WBC) ≥ 3.0×10^9/L; absolute neutrophil count (ANC)≥1.5×10^9/L; hemoglobin≥9.0 g/dL; platelets≥75×10^9/L; serum total bilirubin (TBIL)≤1.5×ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN); serum creatinine≤1×ULN or estimated creatinine clearance ≥ 50 mL/min;
* 6. Left ventricular ejection fraction (LVEF) ≥ 50%;
* 7. Fertile subjects are willing to take contraceptive measures during the study period.
* 8. good compliance and signed informed consent voluntarily

Exclusion Criteria:

* 1. Prior systemic anti-tumor therapy, such as chemotherapy, radiotherapy;
* 2. Participated in other drug clinical trials within 4 weeks;
* 3. History of other malignancies;
* 4. Immunodeficiency, or other immune-related disorders requiring medical intervention;
* 5. Postoperative complications such as bleeding;
* 6. Woman who are pregnant or breastfeeding;
* 7. Drug abuse, or clinical, psychological or social factors that may have an impact on informed consent or the implementation of the study;
* 8.Known allergy to prescription or any component of the prescription used in this study, including nimotuzumab, oxaliplatin, irinotecan, fluorouracil, gemcitabine, and capecitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | Up to 24 months
  The time from the date of surgery to the disease recurrence or death, whichever is earlier.

SECONDARY OUTCOMES:
overall survival (OS) | Up to 24 months
  The time from the date of surgery to death due to any cause.
adverse events | Up to 30 days after last administration
  Frequency and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, MD, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No